CLINICAL TRIAL: NCT00280618
Title: Phase II Study of Eloxatin + 5-Fluorouracil/Leucovorin in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Oxaliplatin in Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L_9202
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin

SUMMARY:
Primary:

* To determine the Tumor Response Rate of patients with hepatocellular carcinoma treated with the combination chemotherapy of Eloxatin+5-Fluorouracil/Leucovorin

Secondary:

* Safety and tolerability of this regimen in these patients

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed hepatocellular carcinoma
* Patients must have measurable disease by CT scan
* Patients with unresectable, recurrent or metastatic disease may be chemonaive or may be previously treated by chemotherapy.
* The period of washout of prior chemotherapy must be greater than 4 weeks from date of randomization. The prior chemotherapy should not include platinum compounds.
* WHO performance status: 0 to 2
* Patients must have adequate organ and marrow function as defined below:

  * Leukocytes : ≥ 3,000/μl
  * Absolute neutrophil count :≥ 1,500/μl
  * Platelets : ≥ 80,000/μl
  * Total bilirubin : < 3.0g/dl
  * ASAT/ALAT : ≤ 3 times the upper normal limits of the institute
  * Creatinine : < 120μmol/l
* Patients with no evidence of clinically significant neuropathy.

Exclusion Criteria:

* Documented allergy to platinum compound or to others study's drugs
* Pregnant or lactating women or women of childbearing potential (e.g. not using adequate contraception)
* Hematological disorder or malignancies
* Metastasis to central nervous system
* Other serious illness or medical conditions:

  * Active infectious disease
  * Congestive heart failure, or angina pectoris. Previous history of myocardial infarction within 1 year from study entry; uncontrolled hypertension or arrhythmia.
* Concurrent treatment with any other anticancer therapy
* Concurrent treatment with other experimental drugs.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-07; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Time to Tumor Progression (TTP) and Response Rate: evaluated by RECIST | During the Study Conduct

SECONDARY OUTCOMES:
Adverse Events collections and evaluation | From the signature of the informed consent up to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Pingkuan Zhang, Study Director — Sanofi